CLINICAL TRIAL: NCT07379996
Title: "Music Therapy in the Recovery Process of Individuals With Severe Mental Disorder in the Community Setting: A Pilot Study."
Brief Title: "Pilot Study of Music Intervention for Recovery of People With Severe Mental Disorder in the Community"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alejando Vargas Rubio (Other)
Responsible Party: Sponsor-Investigator, Alejando Vargas Rubio, Mental Health Nurse Specialist, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CEI.24-93.TFM-A.VargasRubio
Record Dates: First submitted 2026-01-15; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Severe Mental Disorder; Severe Mental Illness
Keywords: Severe Mental Disorder; Hope; Music therapy; Social functioning; Quality of life; Severe mental illness; Mental health recovery; Recovery
MeSH Terms: conditions — Mental Disorders; Social Adjustment

STUDY DESIGN:
Intervention Model Description: Pilot study with a quasi-experimental pre-test and post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with Severe Mental Disorder from an Assertive Community Treatment Team (Experimental): The study was conducted within a community-based service for individuals with Severe Mental Disorder, called the Assertive Community Treatment Team (ACT Team), located in the city of Cartagena, Spain.
  The study participants were active users currently receiving care from this service.
  Interventions: Behavioral: Passive music therapy in an individual format

INTERVENTIONS:
Behavioral: Passive music therapy in an individual format — The intervention was administered individually, and the authors based it on a review of the scientific literature on studies that evaluated the main proposed variables: quality of life, social functioning, and hope.
  In general, participants selected the music they wished to listen to for each session, following the nurse's guidance, and a dialogue was then established between the participant and the nurse.
  The intervention lasted approximately 20 weeks, with a weekly or biweekly frequency. The intervention consisted of 12 sessions, each lasting 45-60 minutes.

SUMMARY:
The aim of this study was to analyze the effect of music therapy on hope, quality of life, and social functioning in individuals with Severe Mental Disorder in the community.

The main research questions were:

Can music therapy increase the level of hope in individuals with Severe Mental Disorder? Can music therapy improve the quality of life of individuals with Severe Mental Disorder? Can music therapy enhance the social functioning of individuals with Severe Mental Disorder?

Participants were users of a Community Mental Health Care Team called the Assertive Community Treatment Team.

A total of 12 music therapy sessions were conducted, each lasting 45-60 minutes. Participants selected the songs or sounds they wanted to listen to based on the session theme, followed by a dialogue between the participant and the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 16 years or older.
* Individuals without severe hearing impairment.
* Individuals without cognitive deficits that would prevent them from reading or understanding the study documents.

Exclusion Criteria:

* Having a severe hearing impairment.
* Inability to read or understand the proposed questionnaires.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF - Quality of Life Scale | This questionnaire was administered at three time points: at baseline (Day 1 of the intervention), at mid-intervention (around Week 10), and at the end of the intervention (Week 20)
  This self-administered questionnaire assesses an individual's quality of life across four domains (physical health, psychological health, social relationships, and environment). It also includes an evaluation of perceived general health and overall quality of life. The questionnaire consists of 26 items with five response options (1-5). The higher the score in each domain, the better the quality of life profile of the person being assessed.
Beck Hopelessness Scale (BHS) | This questionnaire was administered at three time points: at baseline (Day 1 of the intervention), at mid-intervention (around Week 10), and at the end of the intervention (Week 20).
  This self-administered questionnaire assesses an individual's negative perceptions about the future and suicide risk. It consists of 20 items with true/false response options. The results indicate four levels of hopelessness: 0-3 (normal/asymptomatic), 4-8 (mild), 9-14 (moderate), and 15-20 (severe).
Social Functioning Scale (SFS) | This questionnaire was administered at three time points: at baseline (Day 1 of the intervention), at mid-intervention (around Week 10), and at the end of the intervention (Week 20).
  The self-administered version of this scale assesses seven dimensions of social functioning:
  Social isolation: 0 to 3 per item, with a total score range of 0-15. Interpersonal behavior: 4 items. First, items 1 and 2 are summed; if their combined score exceeds 3, a maximum of 3 is assigned. The remaining two items are scored from 0 to 3, resulting in a total score range of 0-9.
  Prosocial activities: 22 items, scored 0 to 3, total score range 0-66. Leisure: 15 items, scored 0 to 3, total score range 0-45. Independence-performance: 13 items, scored 0 to 3, total score range 0-39. Independence-competence: 13 items, scored 1 to 3, total score range 13-39. Employment/occupation: A score of up to 6 points is possible if the patient feels capable of performing some type of work and is making frequent attempts to find employment.
  It includes 78 items. Higher scores consistently indicate a higher level of social functioning in each domain.

SECONDARY OUTCOMES:
Satisfaction with the received intervention | At the end of the intervention, in Week 20.
  The participants completed a self-developed satisfaction survey to assess their level of satisfaction with the intervention, measured using a 5-point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Rehabilitation Unit of Cartagena, Cartagena, Murcia, Spain